CLINICAL TRIAL: NCT00941798
Title: A Randomized, Multi-center, Parallel Group, Double Blind, Study to Assess the Safety of QMF Twisthaler® (500/400 µg) and Mometasone Furoate Twisthaler® (400 µg) in Adolescent and Adult Patients With Persistent Asthma
Brief Title: Safety of QMF149 Twisthaler® in Adolescent and Adult Patients With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQMF149A2210; EudraCT number 2009-011539-10
Record Dates: First submitted 2009-07-14; First posted 2009-07-20 (Estimated); Results first posted 2012-06-05 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Asthma
Keywords: Asthma; LABA; Safety
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- QMF149 Twisthaler® 500/400 (Experimental): QMF149 Twisthaler® (indacaterol maleate 500 µg/mometasone furoate 400 µg), once daily (QD)
  Interventions: Drug: QMF149 Twisthaler®
- Mometasone Twisthaler® (Active Comparator): Mometasone Twisthaler®, 400 µg QD
  Interventions: Drug: Mometasone Twisthaler®

INTERVENTIONS:
Drug: QMF149 Twisthaler® — Once daily via multi-dose dry-powder inhaler
  Arms: QMF149 Twisthaler® 500/400
Drug: Mometasone Twisthaler® — Once daily via multi-dose dry-powder inhaler
  Arms: Mometasone Twisthaler®

SUMMARY:
Study CQMF149A2210 evaluated the safety of QMF149 Twisthaler® 500/400 μg, a fixed dose combination of indacaterol 500 μg, a once daily β2 agonist, and mometasone furoate 400 μg, an inhaled corticosteroid (ICS) that is approved for use in the treatment of asthma. The objective of this safety trial was to assess the effect of treatment on the incidence of serious asthma exacerbations, defined as asthma related hospitalization and/or intubation and/or death. This was an event driven trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented diagnosis of persistent asthma and who were currently treated with or qualified for treatment with both ICS and long-acting beta2-agonist (LABA) combination
* Patients demonstrating an increase in forced expiration volume in 1 second (FEV1) of ≥ 12% or ≥ 200 mLs within 30 minutes after administration of short-acting beta2-agonist (SABA)
* Patients with an FEV1 ≥ 50% of predicted normal

Exclusion Criteria:

* Patients with a previous diagnosis of chronic obstructive pulmonary disease (COPD)
* Patients who had an asthma attack/exacerbation requiring hospitalization/emergency room visit or respiratory tract infection within 1 month prior to randomization
* Patients who had ever required ventilator support for respiratory failure
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Patients with concomitant pulmonary disease
* Patients with certain cardiovascular co-morbid conditions
* Patients with any significant medical condition that might compromise patient safety, interfere with evaluation or preclude completion of the study

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2283 (Actual)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (140):
- United States (86):
  - Novartis Investigator Site, Birmingham, Alabama
  - Novartis Investigator Site, Buena Park, California
  - Novartis Investigator Site, Encinitas, California
  - Novartis Investigator Site, Fullerton, California
  - Novartis Investigator Site, Long Beach, California
  - Novartis Investigator Site, Los Angeles, California
  - Novartis Investigator Site, Orange, California
  - Novartis Investigator Site, Riverside, California
  - Novartis Investigator Site, San Diego, California
  - Novartis Investigator Site, San Jose, California
  - Novartis Investigator Site, San Mateo, California
  - Novartis Investigator Site, Vista, California
  - Novartis Investigator Site, Walnut Creek, California
  - Novartis Investigator Site, Denver, Colorado
  - Novartis Investigator Site, Engelwood, Colorado
  - Novartis Investigator Site, Lakewood, Colorado
  - Novartis Investigator Site, Wheat Ridge, Colorado
  - Novartis Investigator Site, Clearwater, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigator Site, Port Charlotte, Florida
  - Novartis Investigator Site, Sarasota, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigator Site, Tampa, Florida
  - Novartis Investigative Site, Albany, Georgia
  - Novartis Investigative Site, Columbus, Georgia
  - Novartis Investigative Site, Savannah, Georgia
  - Novartis Investigator Site, Couer D'Alene, Idaho
  - Novartis Investigator Site, Chicago, Illinois
  - Novartis Investigator Site, Normal, Illinois
  - Novartis Investigator Site, River Forest, Illinois
  - Novartis Investigator Site, Skokie, Illinois
  - Novartis Investigator Site, Springfield, Illinois
  - Novartis Investigator Site, Evansville, Indiana
  - Novartis Investigator Site, Indianapolis, Indiana
  - Novartis Investigator Site, Iowa City, Iowa
  - Novartis Investigator Site, Topeka, Kansas
  - Novartis Investigator Site, Owensboro, Kentucky
  - Novartis Investigator Site, Metarie, Louisiana
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigator Site, Minneapolis, Minnesota
  - Novartis Investigator Site, Plymouth, Minnesota
  - Novartis Investigator Site, Ozark, Missouri
  - Novartis Investigator Site, Rolla, Missouri
  - Novartis Investigator Site, St Louis, Missouri
  - Novartis Investigator Site, Warrensburg, Missouri
  - Novartis Investigator Site, Bellevue, Nebraska
  - Novartis Investigator Site, Omaha, Nebraska
  - Novartis Investigative Site, Brick, New Jersey
  - Novartis Investigative Site, Cedar Knolls, New Jersey
  - Novartis Investigative Site, Skillman, New Jersey
  - Novartis Investigator Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Mineola, New York
  - Novartis Investigative Site, Newburgh, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative site, Raleigh, North Carolina
  - Novartis Investigator Site, Canton, Ohio
  - Novartis Investigator Site, Columbus, Ohio
  - Novartis Investigator Site, Marion, Ohio
  - Novartis Investigator Site, Sylvania, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigator Site, Oklahoma City, Oklahoma
  - Novartis Investigator Site, Portland, Oregon
  - Novartis Investigative Site, Blue Bell, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigator Site, Lincoln, Rhode Island
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigator Site, Kingsport, Tennessee
  - Novartis Investigator Site, Dallas, Texas
  - Novartis Investigator Site, Dickinson, Texas
  - Novartis Investigator Site, El Paso, Texas
  - Novartis Investigator Site, Fort Worth, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigator Site, Houston, Texas
  - Novartis Investigator Site, New Braunfels, Texas
  - Novartis Investigator Site, San Antonio, Texas
  - Novartis Investigative Site, South Burlington, Vermont
  - Novartis Investigative Site, Abingdon, Virginia
  - Novartis Investigator Site, Kirkland, Washington
  - Novartis Investigator Site, Seattle, Washington
  - Novartis Investigator Site, Tacoma, Washington
  - Novartis Investigator Site, Milwaukee, Wisconsin
- Brazil (6):
  - Novartis Investigative Site, Belo Horizonte
  - Novartis Investigative Site, Florianópolis
  - Novartis Investigative Site, Porto Alegre
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, Salvador
  - Novartis Investigative Site, São Paulo
- Colombia (2):
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
- Czechia (15):
  - Novartis Investigator Site, Boskovice
  - Novartis Investigator Site, Brno
  - Novartis Investigator Site, Brno-Bohunice
  - Novartis Investigator Site, Břeclav
  - Novartis Investigator Site, Hradec Králové
  - Novartis Investigator Site, Jablonec nad Nisou
  - Novartis Investigator Site, Kladno
  - Novartis Investigator Site, Kutná Hora
  - Novartis Investigator Site, Liberec
  - Novartis Investigator Site, Most
  - Novartis Investigator Site, Pilsen
  - Novartis Investigator Site, Prague
  - Novartis Investigator Site, Tábor
  - Novartis Investigator Site, Teplice
  - Novartis Investigative Site, Trutnov
- Hungary (8):
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Debrecen
  - Novartis Investigator Site, Deszk
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Mosonmagyaróvár
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Tatabánya
  - Novartis Investigative Site, Törökbálint
- India (8):
  - Novartis Investigator Site, Chennai
  - Novartis Investigator Site, Coimbatore
  - Novartis Investigator Site, Hyderabaad
  - Novartis Investigator Site, Indore
  - Novartis Investigator Site, Mangalore
  - Novartis Investigator Site, Mumbai
  - Novartis Investigator Site, Nagpur
  - Novartis Investigator Site, Panjim
- Novartis Investigator Site, Lima, Peru
- Slovakia (11):
  - Novartis Investigator Site, Bardejov
  - Novartis Investigative Site, Bojnice
  - Novartis Investigator Site, Bratislava
  - Novartis Investigator Site, Košice
  - Novartis Investigator Site, Levice
  - Novartis Investigator Site, Liptovský Hrádok
  - Novartis Investigator Site, Michalovce
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Šurany
  - Novartis Investigator Site, Trenčín
  - Novartis Investigator Site, Vráble
- South Korea (3):
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative SIte, Seoul
  - Novartis Investigator Site, Seoul

REFERENCES:
- [Derived] Beasley RW, Donohue JF, Mehta R, Nelson HS, Clay M, Moton A, Kim HJ, Hederer BM. Effect of once-daily indacaterol maleate/mometasone furoate on exacerbation risk in adolescent and adult asthma: a double-blind randomised controlled trial. BMJ Open. 2015 Feb 3;5(2):e006131. doi: 10.1136/bmjopen-2014-006131. PMID 25649209

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2283 patients were screened. 1518 patients were randomized.
Period: Overall Study
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Started | 755 | 763
Full Analysis Set | 749 | 759
Completed | 561 | 578
Not Completed | 194 | 185
Not completed — Withdrawal by Subject | 72 | 74
Not completed — Adverse Event | 43 | 23
Not completed — Lost to Follow-up | 29 | 23
Not completed — Protocol Violation | 17 | 20
Not completed — Administrative problems | 13 | 23
Not completed — Lack of Efficacy | 10 | 17
Not completed — Patient's inability to use device | 6 | 1
Not completed — Abnormal test procedure results | 3 | 1
Not completed — Abnormal laboratory values | 1 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler® | Total
Number analyzed (Participants) | 749 | 759 | 1508
Age Continuous [Mean (Standard Deviation); unit: years] | 42.4 (14.75) | 42.3 (14.58) | 42.3 (14.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 436 | 449 | 885
  Male | 313 | 310 | 623

OUTCOME MEASURES:

1. Primary Outcome: Time to First Serious Asthma Exacerbation
Description: Defined as the number of days from start of treatment up to the first date when an asthma exacerbation becomes serious. A serious asthma exacerbation was one that resulted in hospitalization, intubation or death.
Time Frame: Up to 21 months
Population: Full analysis set: all randomized patients who received at least one dose of study medication.
Measure: Median (Full Range); unit: months
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Number analyzed (Participants) | 749 | 759
months | 13.3 [0.0 to 19.6] | 13.4 [0.0 to 20.3]

2. Secondary Outcome: Cumulative Incidence of the First Serious Asthma Exacerbation Resulting in Hospitalization, Intubation or Death.
Description: The number of patients with at least one serious asthma exacerbation over the course of the study. A serious asthma exacerbation was one that resulted in hospitalization, intubation or death.
Time Frame: up to 21 months
Population: Full analysis set: all randomized patients who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Number analyzed (Participants) | 749 | 759
participants | 2 | 6

3. Secondary Outcome: Patients With Asthma Exacerbations That Required Treatment With Systemic Corticosteroids
Description: Number of patients requiring treatment with systemic corticosteroids (oral or parenteral) over the course of the study (up to 21 months).
Time Frame: Up to 21 months
Population: Full analysis set: all randomized patients who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Number analyzed (Participants) | 749 | 759
participants | 124 | 171

4. Secondary Outcome: Number of Patients With at Least One Asthma Worsening Post-baseline
Description: The criterion for asthma worsening were: decrease in peak expiratory flow (PEF) >= 20% from mean baseline on >= 3 consecutive days, nighttime symptom score >= 2 on >= 2 consecutive nights, decrease in forced expiration volume in 1 second (FEV1) >=20% from baseline at evening visits, daytime symptom score of 3 or 4 on >= 2 consecutive days, requiring an urgent unscheduled visit for medical care, 24 hour rescue medication use >= 8 puffs on >= 2 consecutive days, and any other clinically important symptoms (pre-specified MedDRA preferred terms).
Time Frame: Up to 21 months
Population: Full analysis set: all randomized patients who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Number analyzed (Participants) | 749 | 759
participants | 533 | 637

5. Secondary Outcome: Change From Baseline in Trough Forced Expiration Volume in 1 Second (FEV1) at Final Visit
Description: Spirometry was conducted according to internationally accepted standards. Trough FEV1 was measured 15 minutes before dosing; measurements within 6 hours of rescue medication use were set to missing. Repeated measures of analysis of covariance model: change from baseline to trough FEV1 = treatment + visit + treatment*visit interaction + baseline FEV1 + region + asthma related hospitalization in the last 12 months + asthma worsening in the last 12 months + African American patient.
Time Frame: Baseline to the end of treatment (varying durations, up to 21 months)
Population: Full analysis set: all randomized patients who received at least one dose of study medication. Participants with observations at both baseline and final visit were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Number analyzed (Participants) | 674 | 699
liters | 0.06 (0.025) | -0.07 (0.024)

6. Secondary Outcome: Change From Baseline in Forced Expiration Volume in 1 Second (FEV1) at Final Visit
Description: Spirometry was conducted according to internationally accepted standards. Change from baseline at final visit. FEV1 data taken within 6 hours of rescue medication was excluded from the analysis. Repeated measures of analysis of covariance model: change from baseline to final visit FEV1 = treatment + visit + treatment*visit interaction + baseline FEV1 + region + asthma related hospitalization in the last 12 months + asthma worsening in the last 12 months + African American patient.
Time Frame: Baseline to the end of treatment (varying durations, up to 21 months). At the following timepoints: 5 minutes post-dose, 30 minutes post-dose, 1 hour post-dose and 2 hours post-dose
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Number analyzed (Participants) | 578 | 607
liters
  5 minutes post-dose (n = 578, 607) | 0.09 (0.018) | -0.04 (0.018)
  30 minutes post-dose (n = 576, 605) | 0.12 (0.020) | -0.05 (0.020)
  1 hour post-dose (n = 575, 602) | 0.13 (0.021) | -0.06 (0.021)
  2 hours post-dose (n = 568, 601) | 0.14 (0.022) | -0.05 (0.022)

7. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Final Visit
Description: Spirometry was conducted according to internationally accepted standards. Change from baseline at final visit. FVC data taken within 6 hours of rescue medication was excluded from the analysis. Repeated measures of analysis of covariance model: change from baseline to final visit FVC = treatment + visit + treatment*visit interaction + baseline FVC + region + asthma related hospitalization in the last 12 months + asthma worsening in the last 12 months + African American patient.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: liter
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Number analyzed (Participants) | 578 | 607
liter
  5 minutes post-dose (n = 578, 607) | -0.03 (0.023) | -0.11 (0.023)
  30 minutes post-dose (n = 576, 605) | -0.03 (0.025) | -0.13 (0.024)
  1 hour post-dose (n = 575, 602) | -0.01 (0.025) | -0.13 (0.025)
  2 hours post-dose (n = 568, 601) | -0.02 (0.026) | -0.13 (0.026)

8. Secondary Outcome: Changes From Baseline in Morning Peak Expiratory Flow (PEF) and Trough Evening PEF Averaged Over the Entire Post-baseline Period
Description: PEF was performed every morning and evening prior to study medication use except evenings on the day of clinic visits.
  Baseline is average over the last 14 days prior to start of treatment. Analysis of covariance model: change from baseline in PEF = treatment + baseline PEF + region + history of asthma related hospitalization in the past 12 months + history of asthma worsening in the past 12 months + African American patient.
Time Frame: Baseline to the end of treatment (varying durations, up to 21 months)
Population: Full analysis set: all randomized patients who received at least one dose of study medication. Participants with observations at both baseline and at final visit were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: liters per second
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Number analyzed (Participants) | 731 | 748
liters per second
  Morning PEF (n = 730, 746) | 0.43 (0.075) | 0.00 (0.075)
  Evening PEF (n = 731, 748) | 0.27 (0.076) | -0.15 (0.075)

9. Secondary Outcome: Change From Baseline in Percentage of Days With no Asthma Symptoms During the Morning, Daytime and Nighttime
Description: Baseline = the last 14 days prior to start of treatment. Analysis of covariance model: Change from baseline = treatment + baseline value + region + history of asthma related hospitalization in past 12 months + history of asthma worsening in past 12 months + African American patient.
Time Frame: Baseline to the end of treatment (varying durations, up to 21 months)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Number analyzed (Participants) | 731 | 749
percentage of days
  Morning (n = 730, 746) | 22.3 (2.17) | 18.4 (2.17)
  Daytime (n = 731, 749) | 27.1 (2.96) | 19.5 (2.95)
  Nighttime (n = 730, 746) | 23.6 (2.69) | 17.3 (2.68)

10. Secondary Outcome: Change From Baseline in Average Asthma Symptom Score Total, Daytime and Nighttime
Description: Total asthma symptom score = morning symptoms (0, 1) + daytime score (0-4) + nighttime score (0-4). The range is from 0 to 9. A lower number indicates improvement. Baseline = the last 14 days prior to start of treatment.
  Analysis of covariance model: Change from baseline = treatment + baseline value + region + history of asthma related hospitalization in past 12 months + history of asthma worsening in past 12 months + African American patient.
Time Frame: Baseline to the end of treatment (varying durations, up to 21 months)
Population: Full analysis set: all randomized patients who received at least one dose of study medication. Participants with observations at both baseline and endpoint were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Number analyzed (Participants) | 731 | 749
units on a scale
  Total (n = 708, 733) | -1.22 (0.088) | -0.94 (0.088)
  Daytime (n = 731, 749) | -0.50 (0.043) | -0.39 (0.043)
  Nighttime (n = 730, 746) | -0.46 (0.037) | -0.36 (0.037)

11. Secondary Outcome: Change From Baseline in Percentage of Days With no Rescue Medication Use During 24 Hours, Daytime and Nighttime
Description: 24 hours consists of both 12 hour daytime and 12 hour nighttime. Baseline = the last 14 days prior to start of treatment. Analysis of covariance model: Change from baseline = treatment + baseline value + region + history of asthma related hospitalization in past 12 months + history of asthma worsening in past 12 months + African American patient.
Time Frame: Baseline to the end of treatment (varying durations, up to 21 months)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Number analyzed (Participants) | 692 | 711
percentage of days
  24 hours (n = 669, 696) | 29.1 (2.88) | 17.9 (2.88)
  Daytime (n = 692, 711) | 23.6 (2.74) | 13.8 (2.74)
  Nighttime (n = 691, 708) | 24.6 (2.69) | 14.5 (2.68)

12. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) at Final Visit
Description: The Asthma Control Questionnaire score ranges from 0 (good control of asthma) to 6 (poor control of asthma). A negative change in score indicates improvement in asthma control.
  Repeated measures of analysis of covariance model: change from baseline in ACQ score = treatment + visit + treatment*visit interaction + baseline ACQ score + region + asthma related hospitalization in the last 12 months + asthma worsening in the last 12 months + African American patient.
Time Frame: Baseline to the end of treatment (varying durations, up to 21 months)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Number analyzed (Participants) | 675 | 687
units on a scale | -0.55 (0.052) | -0.32 (0.052)

ADVERSE EVENTS:
Arm/Group | QMF149 Twisthaler® 500/400 | Mometasone Twisthaler®
Serious Adverse Events (participants affected / at risk) | 30/749 | 44/759
Other Adverse Events (participants affected / at risk) | 510/749 | 477/759
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QMF149 Twisthaler® 500/400 (N=749) | Mometasone Twisthaler® (N=759)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Chest pain (General disorders) | 1 | 2
Cyst (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 2
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2
External ear cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 4
Septic shock (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Radicular pain (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Colpocele (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Ovarian mass (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QMF149 Twisthaler® 500/400 (N=749) | Mometasone Twisthaler® (N=759)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 | 8
Pyrexia (General disorders) | 9 | 14
Acute sinusitis (Infections and infestations) | 16 | 8
Bronchitis (Infections and infestations) | 39 | 58
Influenza (Infections and infestations) | 26 | 27
Laryngitis (Infections and infestations) | 5 | 12
Lower respiratory tract infection (Infections and infestations) | 13 | 9
Nasopharyngitis (Infections and infestations) | 112 | 106
Pharyngitis (Infections and infestations) | 29 | 27
Respiratory tract infection (Infections and infestations) | 13 | 15
Rhinitis (Infections and infestations) | 21 | 14
Sinusitis (Infections and infestations) | 55 | 52
Upper respiratory tract infection (Infections and infestations) | 83 | 96
Upper respiratory tract infection bacterial (Infections and infestations) | 15 | 21
Urinary tract infection (Infections and infestations) | 14 | 14
Viral infection (Infections and infestations) | 10 | 24
Viral upper respiratory tract infection (Infections and infestations) | 29 | 36
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 11
Headache (Nervous system disorders) | 26 | 30
Asthma (Respiratory, thoracic and mediastinal disorders) | 195 | 269
Cough (Respiratory, thoracic and mediastinal disorders) | 266 | 63
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 | 18
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 29 | 25
Hypertension (Vascular disorders) | 13 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.